CLINICAL TRIAL: NCT04394637
Title: Ultra High Resolution CT to Assess Role of Intramyocardial Fat and Delayed Enhancement in Ventricular Arrhythmogenesis
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00236647
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Arrhythmias
Keywords: Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PROSe-ICD: PROSe-ICD [NCT00733590/ Institutional Review Board (IRB) NA_00045142], a large prospective cohort study of patients who received an ICD for primary prevention.
- Reynolds study: Functional Energetics (Reynolds study, NA_00037404), a study with conventional contrast-enhanced 1H MRI to determine ventricular geometry, global and regional function, as well as infarct size characteristics following delayed contrast enhancement.

SUMMARY:
This research is being done to determine how well cardiac computed tomography (CT) scanning measures of fat within the heart can predict abnormal heart rhythms and how well cardiac CT can measure scar within the heart versus cardiac magnetic resonance imaging (MRI).

* People who have been enrolled in PROSe-ICD (NA_00045142) and Reynolds (NA_00037404) studies may join
* The procedures, tests, drugs or devices that are part of this research and will be paid for by the study

DETAILED DESCRIPTION:
The investigators aim to investigate the role of intramyocardial fat on ventricular arrhythmogenesis. Intramyocardial fat deposition has been frequently observed in patients with ischemic heart disease and is readily detectable by multi-detector computed tomography (MDCT) with high sensitivity and specificity, unlike other modalities. Like intramyocardial fat, reentrant ventricular tachycardia (VT) tends to occur late after the onset of myocardial infarction and the investigators hypothesize that lipomatous metaplasia within the infarct may precipitate later onset ventricular arrhythmias (VA). Prior studies have shown that intramyocardial fat correlates with slow myocardial conduction velocity and with critical circuits for VA but the investigators do not know the causal relationship between intramyocardial fat and future risk of VA.

Intramyocardial fat deposition or lipomatous metaplasia has been frequently observed in patients with ischemic heart disease and is readily detectable by multi-detector computed tomography (MDCT) with high sensitivity and specificity. Like intramyocardial fat, reentrant ventricular tachycardia (VT) tends to occur late after the onset of myocardial infarction and the investigators hypothesize that there may be a causal relationship. Prior studies have shown that intramyocardial fat correlates with slow myocardial conduction velocity and with critical circuits for VT in patients referred for VT ablation who already manifest VA.

However, the correlation of intramyocardial fat on CT with late gadolinium enhancement (LGE) on cardiac magnetic resonance (CMR) in a general population of patients with ischemic cardiomyopathy with no prior history of VA has not been reported. Specifically, it is unknown whether the presence, distribution and/or volume of fat is an independent predictor of VA. Further CMR is less widely available in medical centers, and is more expensive with longer scanning times compared to CT. CT provides higher spatial resolution, is widely available and is not as susceptible to magnetic interference from internal cardiac defibrillator (ICD) generators and thus makes it an attractive imaging modality for risk stratification, particularly longitudinally over time.

Hypothesis: The investigators' objective is to define the prevalence and distribution of intramyocardial fat in patients with ischemic heart disease scheduled for or with in-situ implantable defibrillators. Further, the investigators aim to assess the independent association of intramyocardial fat with VA and determine whether it adds any utility above LGE measured by CMR. Finally, the investigators will assess how well delayed enhanced CT correlates with LGE on MRI and test its association with ventricular arrhythmias.

Importance: The significance of the investigators' research is that the investigators will: 1) test whether intramyocardial fat on CT can be used as a non-invasive tool for sudden cardiac death risk stratification in patients who have or are scheduled to undergo ICDs, and 2) define whether delayed enhancement CT is comparable to the current non-invasive gold standard of CMR for identifying myocardial scar.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older with history of ischemic cardiomyopathy enrolled in the current Reynolds study or PROSe-ICD study will be asked to participate
* Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study CT
* Ability to understand and willingness to sign the Informed Consent Form

Exclusion Criteria:

* Known allergy to iodinated contrast media
* Patients with glomerular filtration rate (GFR) ≤ 30 mL/min will not be enrolled in the study due to the use of intravenous iodinated contrast agents
* Atrial fibrillation or uncontrolled tachyarrhythmia
* Evidence of severe symptomatic heart failure (NYHA Class III or IV)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit patients with a history of an ischemic cardiomyopathy from the current PROSe-ICD to undergo a cardiac CT performed using an ultra-high-resolution (UHR) CT scanner (Canon, Precision) using iodinated contrast for (a) identification of myocardial fat, and (b) myocardial scar visualization (areas of delayed contrast enhancement).
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intramyocardial fat in patients with ischemic heart disease | 2 years
  The primary aim is to test whether intramyocardial fat on MDCT is as effective or adds additional utility to risk stratification for VA above that of CMR-LGE characteristics in ischemic cardiomyopathy patients who are candidates for ICD therapy or have in situ ICDs.
  Our objective is to define the prevalence and distribution of intramyocardial fat in patients with ischemic heart disease scheduled for or with in-situ implantable defibrillators. Further, we aim to assess the independent association of intramyocardial fat with VA and determine whether it adds any utility above LGE measured by CMR.
Prevalence of delayed enhanced CT detected scar | 2 years
  Comparison of the scar distribution on delayed enhanced CT with LGE on cardiac MRI.
  The significance of our research is that we will test whether delayed enhanced CT can be used as a non-invasive tool for sudden cardiac death risk stratification in patients with ischemic heart disease and whether delayed enhancement CT is comparable to the current non-invasive gold standard of CMR for identifying myocardial scar.
Quantification of delayed enhanced CT detected scar | 2 years
  Comparison of the scar distribution on delayed enhanced CT with LGE on cardiac MRI.
  The significance of our research is that we will test whether delayed enhanced CT can be used as a non-invasive tool for sudden cardiac death risk stratification in patients with ischemic heart disease and whether delayed enhancement CT is comparable to the current non-invasive gold standard of CMR for identifying myocardial scar.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chrispin, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No